CLINICAL TRIAL: NCT01271686
Title: 24-hour IOP-lowering Effect of 0.01% Bimatoprost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, John Liu, PhD, Adjunct Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD 101705 bimatoprost
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-05

CONDITIONS: Intraocular Pressure; Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 0.01% bimatoprost (Experimental): bimatoprost 0.01% one time per day at bedtime for 4 weeks.
  Interventions: Drug: 0.01% bimatoprost

INTERVENTIONS:
Drug: 0.01% bimatoprost — 0.01% bimatoprost once in the evening for 4 weeks
  Other Names: Lumigan 0.01%

SUMMARY:
This study will evaluate the 24-hour IOP-lowering efficacy of 0.01% bimatoprost once daily in patients with glaucoma or ocular hypertension

DETAILED DESCRIPTION:
Objectives To investigate the 24 h effects of bimatoprost 0.01% monotherapy on intraocular pressure (IOP) and ocular perfusion pressure (OPP).

Design Prospective, open-label experimental study.

Setting Single tertiary ophthalmic clinic.

Participants Sixteen patients with diagnosed primary open-angle glaucoma (POAG) or ocular hypertension (ages, 49-77 years).

Interventions Baseline data of 24 h IOP in untreated patients were collected in a sleep laboratory. Measurements of IOP were taken using a pneumatonometer every 2 h in the sitting and supine body positions during the 16 h diurnal/wake period and in the supine position during the 8 h nocturnal/sleep period. After baseline measurements were taken, patients were treated with bimatoprost 0.01% one time per day at bedtime for 4 weeks, and then 24 h IOP data were collected under the same laboratory conditions.

Primary outcome measure of nocturnal IOP mean under bimatoprost 0.01% treatment was compared with baseline.

ELIGIBILITY:
Inclusion Criteria:

* primary open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* Women of childbearing potential previous glaucoma surgery presence of other eye disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Liu, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Shiley Eye Center, La Jolla, California, United States

REFERENCES:
- [Result] Tung JD, Tafreshi A, Weinreb RN, Slight JR, Medeiros FA, Liu JH. Twenty-four-hour effects of bimatoprost 0.01% monotherapy on intraocular pressure and ocular perfusion pressure. BMJ Open. 2012 Aug 23;2(4):e001106. doi: 10.1136/bmjopen-2012-001106. Print 2012. PMID 22918671
- See also: Open access publication — http://bmjopen.bmj.com/content/2/4/e001106.full

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Experimental subjects were recruited consecutively from patients with diagnosed bilateral primary open angle glaucoma or ocular hypertension at the Hamilton Glaucoma Center of the University of California, San Diego.
Pre-assignment Details: Subjects who smoked, had previous glaucoma surgery in either eye, had a history of ocular trauma or a sleep disorder, or had an irregular sleep schedule were excluded.
Groups:
- 0.01% Bimatoprost: 0.01% bimatoprost: 0.01% bimatoprost eye drop once in the evening both eyes for 4 weeks
Period: Overall Study
Arm/Group | 0.01% Bimatoprost
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 0.01% Bimatoprost
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Nocturnal Intraocular Pressure (IOP) Change
Description: Nocturnal IOP means under bimatoprost 0.01% treatment were compared with baseline.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 0.01% Bimatoprost
Number analyzed (Participants) | 16
mmHg | -2.6 (2.8)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | 0.01% Bimatoprost
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No